CLINICAL TRIAL: NCT01873911
Title: Characterizing the Neurobehavioral Phenotype(s) in MPS III
Brief Title: Neurobehavioral Phenotypes in MPS III
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National MPS Society (Other); Shire Human Genetic Therapies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0806M35341; U54NS065768 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-06-10 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sanfilippo Syndrome Type A; Sanfilippo Syndrome Type B; Hurler Syndrome
Keywords: MPS IIIA; MPS IIIB; Sanfilippo syndrome type A; Sanfilippo syndrome type B; Hurler syndrome; cognitive decline; MPS IH
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidosis I; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothesis #1: Factor analysis of the revised Sanfilippo Behavior Rating Scale (SBRS) will identify a group of externalizing behaviors and a group of Klüver-Bucy syndrome-like behaviors as two different factors that are at least partially independent.

Hypothesis #2a: Children with MPS III will show more hyperlocomotion, fearlessness, asociality and noncompliance than children of similar cognitive ability with MPS I.

Hypothesis #2b: These behaviors will become more frequent and/or intensify over time, consistent with the Cleary and Wraith (1993) model. Quantifying them will provide a more empirical framework for staging disease progression.

Hypothesis #3: Brain volumetric analysis and diffusion-tensor imaging will reveal abnormalities of frontal and temporal lobe structures that will correlate with externalizing and Klüver-Bucy syndrome-like behaviors, respectively.

Hypothesis #4. Loss of cognitive and language function as measures of neurologic decline will directly precede or co-vary with behavioral decline.

The primary objective of this study is to identify the behavioral phenotype and its neural basis in MPS III (Sanfilippo syndrome). Is the behavioral phenotype similar to that of Klüver-Bucy syndrome, and is there evidence for amygdala abnormality? The secondary objective of this research study is to develop easily administered, sensitive and specific neurobehavioral and neuroimaging markers to characterize the behavioral phenotype(s) of MPS III; to track their progression; and to delineate their neural substrates. Such markers are critical for identifying the stage of disease for each patient, and to measure treatment outcome. Although we know that severe cognitive decline is one essential characteristic of MPS III, the other highly salient characteristic is a range of abnormal and disruptive behaviors that can include, but go well beyond, childhood noncompliance and oppositionality. These behaviors set Sanfilippo syndrome apart from the other MPS disorders. They cause major disruption in the child's familial, school, and community environments. Delineating these behavioral abnormalities will help in better understanding the neurological disease.

DETAILED DESCRIPTION:
Like some other mucopolysaccharidosis (MPS) syndromes, MPS III (Sanfilippo syndrome) is characterized by a severe cognitive decline ending in dementia and death. Unlike other MPS syndromes, earlier-stage MPS III is also associated with a range of abnormal and disruptive behaviors that can include, but go well beyond, childhood noncompliance and oppositionality. These behaviors, which cause major disruption in the child's familial, school, and community environments, set MPS III apart from the other MPS disorders. These behaviors may also indicate the identity of the neural pathways affected in this disease; their sequence of onsets may indicate the order in which these pathways are affected. We propose to define and categorize the behavioral profile(s) or phenotype(s) of MPS III and correlate them with clinical quantitative neuroimaging in order to understand the neural bases of the disease. In addition, we will use these results to develop a set of sensitive and specific measures that can be easily administered by health care professionals to help monitor the disease and the efficacy of future treatments.

ELIGIBILITY:
Inclusion Criteria:

Research Subjects: Verified diagnosis of MPS IIIA or MPS IIIB (having proof of either genetic mutation or enzymatic analysis prior to enrollment in this study); must be between the ages of 2 and 12 years; must be able to walk.

Control group: Verified diagnosis of MPS IH; must have already undergone hematopoietic cell transplantation in the past; must be aged between 2 and 5 years; and must be able to walk without support.

Exclusion Criteria:

Participants will be excluded who are unable to cooperate or comply with this study's procedures; in the opinion of the principal investigator, participants who have other severely-limiting co-existing conditions such as severe hearing or visual impairment, will be excluded from this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twenty children who have been diagnosed with MPS III type A or type B. Ten age-matched children (as controls) who have been diagnosed with MPS I (Hurler syndrome), who in the past have undergone hematopoietic cell transplantation, and who have been clinically-determined to have low cognitive function.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Temperament | Within One Year of Enrollment
  Using Risk Room procedures of the established "Laboratory Temperament Assessment Battery" (Lab-TAB), the investigators will measure and record each subject's startle, exploration (fear), compliance, and attachment.

SECONDARY OUTCOMES:
Quality of Life Measures | Within One Year of Enrollment
  Assessments of research subjects' quality of life will be made using age-appropriate standardized assessment tools.
Event-Related Potentials Measurement | Within One Year of Enrollment
  High-density Event-Related Potentials (ERPs) will be elicited and recorded. ERPs provide information about the timing and location of neurocognitive processes associated with the individual's processing of discrete stimuli. Two sets of stimuli will be used: 1. auditory stimuli consisting of non-language sounds and phonemes; and 2. visual stimuli consisting of images of emotional faces. All stimuli will be presented in an oddball paradigm format (repetition of stimuli with a random insertion of a novel stimulus).
Magnetic Resonance Imaging Examination | Within One Year of Enrollment
  To examine the neural substrate of MPS III behavioral phenotypes of participating research subjects, the investigators will perform high-resolution brain volumetric magnetic resonance imaging (MRI) during clinical scans.
Assessment of Cognitive Development | Within One Year of Enrollment
  Research subjects' cognitive development will be assessed using age-appropriate standardized assessment tools.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa G Shapiro, PhD, Principal Investigator — University of Minnesota; Michael Potegal, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Cleary MA, Wraith JE. Management of mucopolysaccharidosis type III. Arch Dis Child. 1993 Sep;69(3):403-6. doi: 10.1136/adc.69.3.403. No abstract available. PMID 8215557
- [Background] Meyer A, Kossow K, Gal A, Muhlhausen C, Ullrich K, Braulke T, Muschol N. Scoring evaluation of the natural course of mucopolysaccharidosis type IIIA (Sanfilippo syndrome type A). Pediatrics. 2007 Nov;120(5):e1255-61. doi: 10.1542/peds.2007-0282. Epub 2007 Oct 15. PMID 17938166
- [Background] Jha S, Patel R. Kluver-Bucy syndrome -- an experience with six cases. Neurol India. 2004 Sep;52(3):369-71. PMID 15472430
- [Background] Angrilli A, Mauri A, Palomba D, Flor H, Birbaumer N, Sartori G, di Paola F. Startle reflex and emotion modulation impairment after a right amygdala lesion. Brain. 1996 Dec;119 ( Pt 6):1991-2000. doi: 10.1093/brain/119.6.1991. PMID 9010003
- See also: National MPS Society — http://www.mpssociety.org/